CLINICAL TRIAL: NCT03000556
Title: 0.3% Sodium Hyaluronate Eye Drop to Prevent Recurrent Corneal Epithelium Exfoliation After Corneal Abrasions: a Pilot Study
Brief Title: 0.3% Sodium Hyaluronate Eye Drop to Prevent Recurrent Corneal Epithelium Exfoliation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fang Duan (Other)
Responsible Party: Sponsor-Investigator, Fang Duan, clinical professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AL-2016-DF
Record Dates: First submitted 2016-12-14; First posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Corneal Epithelium Exfoliation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experience (Experimental)
  Interventions: Drug: 0.3% Sodium Hyaluronate Eye Drop
- control (No Intervention)

INTERVENTIONS:
Drug: 0.3% Sodium Hyaluronate Eye Drop — The patients need to use 0.3% Sodium Hyaluronate Eye Drop for 3 month.
  Arms: experience

SUMMARY:
Corneal abrasion (TCA) is the most common ophthalmic emergency disease, accounting for about 10% of the American ophthalmic emergency, accounting for 22% of the ophthalmic emergency in Zhongshan Ophthalmic Center. Clinical emergency treatment of TCA is relatively simple and effective, corneal epithelial damage can be recovered within 48 hours. However, about 25% TCA would be developed to the recurrence of exfoliation. Once the recurrence of TCA, the treatment would be more difficult and even cause blindness. Therefore, it is of great practical significance to prevent the recurrence of TCA. However, there is no effective methods to prevent recurrence of TCA.

0.3% sodium hyaluronate eye drops can effectively supplement the shortage of tear and promote repair of corneal epithelium. On this basis, the investigators hypotheses that 0.3% sodium hyaluronate eye drops can prevent the recurrence of TCA. So, investigators intend to test effectiveness of 0.3% sodium hyaluronate drops to prevent the recurrence of TCA by a prospective, single center, randomized, controlled pilot study. In this study, 60 patients with TCA were randomly divided into control group and sodium hyaluronate treatment group and observed one year.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of primary corneal epithelial abrasion;
* Monocular onset;
* Corneal epithelium was defected and fluorescein sodium staining was positive.

Exclusion Criteria:

* Corneal epithelial defect complicated with infection
* Associated with other ocular surface disease patients (such as hypophasis, meibomian gland dysfunction, keratoconjunctivitis sicca syndrome, bullous keratopathy, corneal dystrophy and drug-induced corneal toxicity etc.)
* Pregnant or lactating women; serious heart, liver, and kidney dysfunction; mental disorders; other inflammatory or autoimmune diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of recurrent corneal epithelium exfoliation | 6 month
  Recurrent corneal epithelial exfoliation was defined as positive staining of corneal fluorescein by slit lamp microscope and the patient had obvious eye pain.

SECONDARY OUTCOMES:
the incidence of recurrent corneal epithelium exfoliation | 1 year
  Recurrent corneal epithelial exfoliation was defined as positive staining of corneal fluorescein by slit lamp microscope and the patient had obvious eye pain.
corneal fluorescein staining score | 1 year
  Grading of corneal epithelial fluorescein sodium staining under slit lamp. The average cornea was divided into four quadrants and scored separately, adding all the scores to get the final score. Scoring criteria: 0 point: no staining; 1 point: punctate staining less than 30 dots; 2 points: punctate staining more than 30 dots, more than the point of the color but not scattered; 3 points: severe dispersion staining but no plaque staining; 4 points: plaque staining. Maximum score of 16 points per eye.
Corneal edema grading | 1 year
  Grading of corneal edema under slit lamp. 0 point: C、corneal transparency without edema; 1 point: corneal haze edema, corneal endothelium smooth, iris texture is clearly visible; 2 points: corneal surface roughness, iris texture fuzzy; 3 points: corneal endothelial surface cracking, iris texture as is not clear; 4 points: white corneal edema, intraocular structure as unclear.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan ophthalmic center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wei M, Zou Y, Duan F, Ding X, Zhuang J, Deng J, Yuan Z. Efficacy of Long-term Use of 0.3% Sodium Hyaluronate Eye Drops for Traumatic Corneal Abrasion: A Randomized Controlled, Pilot Trial. Cornea. 2021 Oct 1;40(10):1248-1252. doi: 10.1097/ICO.0000000000002625. PMID 33369934